CLINICAL TRIAL: NCT01001390
Title: The Effects of Ankle Foot Orthoses on Gait Efficiency in Children With Acute Lymphoblastic Leukemia and Foot Drop
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study closed due to poor accrual and difficulty with participant compliance.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GAIT09
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-01

CONDITIONS: Foot Drop; Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic leukemia
MeSH Terms: conditions — Peroneal Neuropathies; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group One (Other): Group one will take a six minute walk test with AFO device, and after a rest of fifteen minutes, they will take another six minute walk test without AFO, with similar speed to the previous test.
  Interventions: Device: AFO Device
- Group Two (Other): Group two will take a six minute walk test without AFO device, and after a rest of fifteen minutes, they will take another six minute walk test with AFO, with similar speed to the previous test.
  Interventions: Device: AFO Device

INTERVENTIONS:
Device: AFO Device — Ankle Foot Orthoses impact on net oxygen consumption.

SUMMARY:
This study is designed to see if children with acute lymphoblastic leukemia who have developed foot drop during treatment for their leukemia consume less oxygen when walking with or without an ankle brace designed to support their foot during walking. In this study children with foot drop are asked to walk for six minutes with and without brace on their ankle. During each walk, the amount of oxygen used is measured. The child wears a face mask which is attached to a device that records how much oxygen they use. The amount of oxygen used during the walk with the brace on will be compared to the amount of oxygen used with the brace off.

DETAILED DESCRIPTION:
1. This study will determine the impact of Ankle Foot Orthoses (AFO) wear on gait efficiency in children with ALL and Chemotherapy-Induced Peripheral Neuropathy (CIPN).
2. The study hypothesizes that children with CIPN will have lower net oxygen consumption during the six minute walk test while wearing AFO as compared to their net oxygen consumption during a six minute walk test while not wearing AFO.
3. The study will assess whether gait efficiency while using an AFO persists after one month of use.
4. The study will hypothesize that the benefits of AFO use on gait efficiency persist after one month of wear.

ELIGIBILITY:
Inclusion Criteria:

1. Research participant is diagnosed with childhood ALL and currently being treated on the TOTAL XVI protocol at St. Jude Children's Research Hospital (SJCRH)
2. Research participant is from 6 to 18 years of age at the time of the scheduled evaluation
3. Research participant has chemotherapy-induced peripheral neuropathy resulting in foot drop
4. Research participant will be receiving AFO
5. Research participant has a hemoglobin level greater than 8 g/dL and a platelet count above 50 x 109/L

Exclusion Criteria:

1. Participant has Down Syndrome or other known congenital developmental delays
2. Participant has a platelet count lower than 50 x 109/L and a hemoglobin level less than 8 g/dL
3. Participant has a lower extremity amputation, congenital deformity of the lower limb or an acute fracture of the lower limb
4. Participant has symptomatic osteonecrosis in the lower extremities

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K Ness, PT, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants were enrolled at St. Jude Children's Research Hospital (SJCRH) between February 2010 and January 2011. The study was terminated due to poor accrual and poor participant compliance.
Pre-assignment Details: Participants had a diagnosis of acute lymphoblastic leukemia and had developed foot drop during treatment for their leukemia. Randomization was to one of two reporting groups: (1) With then without AFO, and (2) Without then with AFO.
Groups:
- Group 1: With Then Without AFO: Group one participants were to complete a six minute walk test with ankle foot orthoses (AFO), and after a rest of fifteen minutes, they were to complete another six minute walk test without AFO, with similar speed to the previous test. The process was to be repeated one month later.
- Group 2: Without Then With AFO: Group two participants were to complete a six minute walk test without ankle foot orthoses (AFO), and after a rest of fifteen minutes, they were to complete another six minute walk test with AFO, with similar speed to the previous test. The process was to be repeated one month later.
Period: Overall Study
Arm/Group | Group 1: With Then Without AFO | Group 2: Without Then With AFO
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Failure to wear AFO device | 2 | 0

BASELINE CHARACTERISTICS:
Population: Two participants were enrolled, however, neither participant continued to wear their ankle foot orthoses after the initial visit.
Arm/Group | Group 1: With Then Without AFO
Number analyzed (Participants) | 2
Age, Customized [Number; unit: participants]
  < 6 years | 0
  6-18 years | 2
  > 18 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Net Oxygen Consumption During the Six Minute Walk Test Among Study Participants Under the Two Walking Conditions, With and Without AFO.
Description: Net oxygen consumption is calculated by the formula: [net oxygen consumption = walking oxygen consumption - sitting oxygen consumption], then adjusted by total mass in kg, including body mass, the mass of the socks, appropriate shoes, helmet, mouth piece system, and for the with AFO trials, the mass of the brace.
Time Frame: Baseline
Population: No data was collected for analysis. Two participants were enrolled, however, neither participant agreed to wear an ankle foot orthoses.
Arm/Group | Group 1: With Then Without AFO
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Improvement in Gait Efficiency While Using an AFO
Description: The difference of net oxygen consumption between wearing AFO and without wearing AFO (difference = wearing AFO - without wearing AFO) will be compared between the baseline study and one month later by using repeated measures analysis in which the effect of time will be tested controlling for other confounding variables.
Time Frame: One month after baseline evaluation
Population: as for outcome 1
Arm/Group | Group 1: With Then Without AFO
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were to be monitored for possible adverse events from the time of enrollment through the six-month follow-up testing. The study terminated early, and no adverse events were experienced.
Description: Two participants were enrolled in Group 1 (With Then Without AFO). No participants were enrolled in Group 2 (Without Then With AFO).
Arm/Group | Group 1: With Then Without AFO | Group 2: Without Then With AFO
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated due to poor accrual and poor participant compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes